CLINICAL TRIAL: NCT05676736
Title: Impact of Obesity on Periodontal Health in a Sample of Adult Egyptian Patients: A Comparant Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Zakaria Ibrahium Mohammed, Associate professor Oral Medicine & Periodontology, Cairo University
Other Study IDs: Mai Zakaria Protocol
Record Dates: First submitted 2022-12-31; First posted 2023-01-09 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Obesity, Periodontal Health
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group (S) Obese group: Patients with body mass index (BMI) range from (≥30 kg/m2)
  Interventions: Other: No intervention
- Control group (C) Normal weight group: Patients with body mass index (BMI) range from (18.5-24.9 kg/m2)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention to be done for the group

SUMMARY:
Periodontal disease is deﬁned as "an inﬂammatory disease of the tooth supportive structure caused by speciﬁc microorganisms or groups of speciﬁc microorganisms, resulting in progressive destruction of the periodontal ligament and alveolar bone with increased probing depth formation, recession, or both". According to WHO, overweight and obesity are defined as abnormal or excessive fat accumulation that may impair health. Body mass index (BMI) can be considered as an indicator of obesity-related health risks. Obesity was considered a global epidemic problem by the World Health Organization in the 1990s as it has increased internationally over the last decades. Based on review in 2003 the periodontal disease onset, progression and response to therapeutic interventions have been shown to be inﬂuenced by several systemic, local and environmental modifying factors and the data collected from the literature suggests that nutritional supplementation has been suggested as a possible inﬂuencing factor on periodontal status and wound healing.

DETAILED DESCRIPTION:
* Dental patients will be recruited in a consecutive manner from the outpatient Diagnostic center, Faculty of Dentistry, Cairo University.
* To estimate the level of overweight and obesity. commonly used the (BMI); was calculated as the body weight (kg) divided by the square of the height (m).
* A total number of 384 patients will be included in this study. The patient categorized as obese will serve as study group (S group) and the patients categorized as normal weight patients will serve as control group (C group).
* Medical history will be taken, thorough oral examination will be done, and a full questionnaire will be filled for each patient.
* Before filling the questionnaire, the aim of the study will be explained to the patient and the patient's acceptance to participate in the survey will be received.
* Non-respondent patients or patients refusing to participate will be reported with the cause of their refusal.
* The questionnaire will be filled through a face-to-face personal interview with the patient using simple, short, easily comprehended questions.
* Full questionnaire will be filled, then full mouth periodontal examination and charting will be done for each patient.
* The interview questions will be prepared in English, translated into Arabic and then reverse translated by a certified translator to ensure accuracy.
* All the interviews will be done by the same investigator.
* Clinical examination will be held on a dental unit using the light of the unit and a mirror. Periodontal health status will be evaluated by full mouth charting using UNC 15 periodontal probe, including assessment of Probing Depth (PD), Clinical Attachment Level (CAL), Bleeding on probing (BOP), plaque index (PI), body mass index (BMI) and health eating index (HEI).
* The questionnaire which was applied in study will include the following:
* Questions including section for demographic information of age, gender, marital status, income, weight, length.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age is between 18-60 years old.
2. Provide informed consent.
3. Patient have at least 20 natural teeth.
4. Patient had no received periodontal treatment within previous 4 months.

Exclusion Criteria:

1. Individuals with chronic systemic diseases such as cancer, osteoporosis, endocrine and hematological Pathologies.
2. Patients having problem in opening their mouth or undergoing intermaxillary fixation where oral examination will not be possible.
3. Pregnant women.
4. Patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs.
5. Patients with orthodontic appliances.
6. Patient had autoimmune condition.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: - Dental patients will be recruited in a consecutive manner from the outpatient Diagnostic center, Faculty of Dentistry, Cairo University.
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
- The primary outcome of the study is the periodontal health in association with obesity | Day 1
  The periodontal health status evaluated by full mouth charting using UNC 15 peiodontal probe, including probing depth (PD), clinical attachment Level (CAL), bleeding on probing (BOP), plaque index (PI).

CONTACTS AND LOCATIONS:
Overall Officials: Mai Zakaria, ph, Principal Investigator — Associate professor Oral Medicine & Periodontology, Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
individual participant data are not to be shared with other researchers until publication of the study.